CLINICAL TRIAL: NCT03058094
Title: A Phase III, Open-Label, Randomized Multicenter Study to Compare AC0010 and Pemetrexed/Cisplatin in Patients With Advanced NSCLC Who Have Progressed Following Prior EGFR TKI
Brief Title: A Study Comparing AC0010 and Chemotherapy in Patients With Advanced NSCLC Who Have Progressed Following Prior EGFR TKI
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Considiering to change the Chemotherapy into Gefitinib
Sponsor: Hangzhou ACEA Pharmaceutical Research Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AEGIS2:AC201602AVTN04
Record Dates: First submitted 2016-12-01; First posted 2017-02-20 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: NSCLC
MeSH Terms: interventions — Pemetrexed; Cisplatin; abivertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AC0010 (Experimental): AC0010, 300mg, orally, BID with a 21-day cycle
  Interventions: Drug: AC0010
- Chemotherapy (Active Comparator): pemetrexed 500 mg/m2 + cisplatin 75 mg/m2 on day one of 21-day cycle, with total of 4-6 cycles.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin 75mg/m2

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed will be administered as an intravenous infusion over 10 minutes on Day 1 of each 21-day cycle. Folic acid will be administered 1-2 weeks prior to the 1st dose, then daily during the treatment period until 21days post the last dose. Vitamin B12 will be administered on the same day of pemetrexed infusion during the treatment period. Corticosteroid will be adminstered on the day prior to, on the day, and on the day after infusion.
  Other Names: Alimta
  Arms: Chemotherapy
Drug: Cisplatin 75mg/m2 — Cisplatin will be administered as an intravenous infusion.
  Other Names: cis-platinum
  Arms: Chemotherapy
Drug: AC0010 — 300mg, orally, BID
  Other Names: AC0010MA
  Arms: AC0010

SUMMARY:
A Phase III, Open-Label, Randomized Multicenter Study to Compare AC0010 and Pemetrexed/Cisplatin in Patients With Advanced NSCLC Who Have Progressed Following Prior EGFR TKI.

DETAILED DESCRIPTION:
This is a phase III, open label, randomized study assessing AC0010 (300 mg, BID) versus pemetrexed/cisplatin (4-6 cycles) in patients with advanced NSCLC, who have progressed following prior therapy with EGFR-TKI.

Patients must provide a biopsy for central confirmation of T790M mutation positive. Eligible patients will be randomized (2:1) into AC0010 group or pemetrexed/cisplatin group. Patients in chemotherapy group can cross-over to AC0010 treatment when patients experience disease progression or intolerability of chemotherapy. The primary objective of the study is to compare the PFS of AC0010 and pemetrexed/cisplatin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18-75 years old.
2. Histological or cytological confirmed diagnosis of locally or metastatic NSCLC (stage IIIB/IV).
3. Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy.
4. Radiological proven disease progression while on first generation EGFR TKIs.
5. At least one measurable disease according to RECIST 1.1.
6. Confirmation of tumor EGFR sensitive mutation positive in previous tumor samples, including G719X, exon 19 deletion, L858R, L861Q.
7. Confirmation of tumor harboring of T790M mutation by central lab with a biopsy sample taken after failure of first generation EGFR TKIs.
8. Adequate organ function:

   * Bone marrow reserve: Absolute neutrophil count ≥1.5 ´ 109/L,. Platelet count ≥100´ 109/L , Hemoglobin≥9 g/dL
   * Liver function: Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤2.5 × the upper limit of normal (ULN) or <5 times ULN in the presence of liver metastases; Total bilirubin ≤1.5 × ULN
   * Kidney function: Creatinine ≤1.5 × ULN
9. Anti-cancer treatment prior to EGFR TKIs including chemotherapy, radiotherapy and other anti-cancer drugs for advanced stage is not allowed.
10. Resolved toxicities from prior therapy less than CTCAE grade 1 (except alopecia) and minimum 7 days of washout period from previous erlotinib, gefitinib or icotinib.
11. ECOG performance status 0 to1.
12. Life expectancy more than 3 months.
13. Patients without CNS metastases or asymptomatic patients with brain metastases. End of local therapy for brain metastases, including radiotherapy and surgery is required ≥28 days prior to beginning of screening.
14. Provision of signed informed consent.

Exclusion Criteria:

1. Undiagnosed by pathology.
2. HCV antibody positive, active hepatitis B (hepatitis B virus carrier can be recruited)
3. HIV antibody positive, other acquired immunodeficiency disease and congenital immunodeficiency disease. Patients with organ transplantation.
4. Patients received new aided/aided system therapy with palindromia in 12 months, the new aided/aieded system therapy is considered to be previous first-line treatment.
5. Condition of organ system:

   * Large field radiation or radiation field covered more than 30% bone marrow within 4 weeks of enrollment.
   * A past history of interstitial lung disease, drug-induced interstitial lung disease or other active interstitial lung disease with clinical proof
   * Idiopathic pulmonary fibrosis (IPF).
   * In the investigator opinion, any severe or uncontrolled disease, such as unstable or uncontrolled respiratory, cardiovascular, liver or kidney diseases.
   * Any unstable system disease including refractory hypertension, unstable angina pectoris, congestive heart-failure, liver and renal disease, metabolic disease.
   * Patients with other malignant tumor in 5 years (except cured cervical carcinoma in situ, Basal cell carcinomas, squamous cell carcinoma)
   * A past history of neurological disorder or mental disorder including epilepsy and dementia.
   * Patients with chronic gastrointestinal diseases, inability to swallow medication, malabsorption syndrome or previous significant bowel resection that would preclude adequate absorption of AC0010.
6. Uncontrolled pleural and pericardial effusion.
7. Patients who have used high-dose glucocorticoids or other immunosuppressive agents within 1 month prior to screening.
8. Patient with symptomatic CNS metastases.
9. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 6 months, heart block with second degree or greater, QTcB > 430ms（male）or > 450ms（female）.
10. Patients receiving medication known to prolong QT interval and potent inducers and inhibitors of CYP3A4 within 4 weeks of fist dose of AC0010.
11. Patients prove 1ml plasma to site's central lab after signing informed consent and the test results show the medication of AZD9291.
12. Patients who have been registered and received the study treatment or withdrawn from the study cannot be enrolled.
13. Patients receive unrelated surgery more than 14 days prior to the screening.
14. Pregnant and lactating women.
15. Women with childbearing potential are defined as all women who are physiologically able to have a pregnancy, unless they are using an efficient contraceptive method during treatment and within 7 days after discontinuation of treatment.
16. Men who have sexual intercourse unless they use a condom during sexual intercourse during treatment and 7 days after discontinuation of treatment and do not impregnate their sexual partners during the period. Vasectomized males are also required to use condoms to prevent the transmission of drugs through semen.
17. Patients who are considered by the investigator as inappropriate to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of randomization until the date of first documented progression or the date of death from any cause, whichever came first, assessed up to 24 months.
  To assess the Progression-Free Survival (PFS) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline up to 28 days after completion of study drug, assessed up to 24 months.
  To assess the overall objective response rate (ORR) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
Duration of Response (DoR) | From occurring of CR or PR until progression or the date of death from any cause, whichever came first, assessed up to 24 months.
  To assess the overall objective response rate (ORR) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
Disease Control Rate (DCR) | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  To assess the Disease Control Rate (DCR) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
Overall Survival (OS) | From the date of randomization to death or end of study, which is assessed up to 36 months.
  To assess the Overall Survival (OS) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
Patient Reported Outcomes by EORTC QLQ-C30 Questionnaire | Baseline up to 28 days after completion of study drug, assessed up to 24 months.
  To assess the safety of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).

OTHER OUTCOMES:
Incidence of toxicity, grading with CTCAE 4.03 | From the date of randomization until end of treatment,which is assessed up to 24 months
  Clinical chemistry, hematology, urinalysis, vital signs, physical examination, weight, ECG and ECOG Performance status and adverse event will be used to assess safety endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (21):
- China (21):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese General PLA Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital Army Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fuzhou General Hospital of Nanjing Military Command, Fuzhou, Fujian
  - Tumor Hospital of Hebei Province, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing General Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital & Institute, Chengdu, Sichuan
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital,Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No